CLINICAL TRIAL: NCT00296920
Title: Deep Brain Stimulation for Refractory Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-0118-B
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2005-09

CONDITIONS: Major Depressive Disorder
Keywords: Deep Brain Stimulation; Treatment failure
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation

SUMMARY:
Despite many available treatments, there are patients with major depression who remain treatment refractory and chronically disabled. For these severely ill patients, several neurosurgical procedures are available where brain lesions are made that interrupt white matter tracts linking orbital frontal cortex to the striatum, resulting in significant therapeutic benefit for many patients. In this study, we will test the safety and efficacy of Deep Brain Stimulation (DBS)--a reversible method used to modulate brain activity--as an alternative to the standard subcaudate tractotomy (SCT). The physiological consequences of this procedure will be mapped longitudinally using positron emission tomography (PET) measures of brain glucose metabolism. Patients will be clinically monitored for 1 year with longitudinal psychiatric, neurological, neurosurgical, neuropsychological and PET imaging examinations to assess treatment efficacy and side effects.

DETAILED DESCRIPTION:
Study Design Subjects: Ten patients will be enrolled in this pilot study. Eligibility criteria: (i) age 30-70 years old, (ii) diagnosis of refractory unipolar major depression, (iii) recurrent illness with a minimum four major depressive episodes, (iv) current episode duration of no less than twelve months; (v) current episode treatment failure to a minimum of four treatment classes-including serotonin-reuptake inhibitors (SSRI), other novel agents, monoamine oxidase inhibitors (MAOI), tricyclics; somatic treatments such as ECT or vagus nerve stimulation (VNS); some form of psychotherapy. Exclusion criteria (i) previous brain surgery (ii) neurological disorder of any type, (iii) significant psychiatric comorbidity as defined by DSM IV diagnostic criteria (such as schizophrenia, panic disorder) (iv) serious medical conditions or contraindication for surgery such as cardiac pacemaker/defibrillator or other implanted devices. Full medical records from a treating psychiatrist will first be reviewed by Dr. Kennedy. Eligible patients will then undergo a full psychiatric, neurological and neuropsychological evaluation (Appendix 1 and 2). Final selection will be made by consensus of the investigative team in collaboration with a senior independent psychiatrist Robert Cooke, MD with expertise in intractable mood disorders. Informed consent will be obtained prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70; men and women (non-pregnant)
* Diagnosis: major depressive episode (unipolar) by DSM-IV derived from the SCID-P.
* Recurrent disease; minimum 4 major depressive episodes .
* Chronic illness with current episode ~ 12 months duration
* Response failure to multiple treatment regimens. Resistance or intolerance to at least four treatments from different categories (SSRI, SNRI, TCA, HCA, MAOI, atypical, Lithium, anticonvulsants, ECT, VNS, CBT/IPT). Documentation of adequate dose and duration of each treatment.
* Hamilton Rating Scale for Depression (HRSD-24) score >20
* Global Assessment of Function. score ~50
* No neurological disease; no other Axis 1 or Axis II diagnosis; no substance abuse
* Stable on current antidepressant meditation regimen or medication free ~4 weeks
* Able to give informed consent in accordance with institutional policies.
* Able to comply with all testing and follow-up visit requirements defined by the Study Protocol. Pre-menopausal women must agree to use acceptable methods of birth control (radiation risk of PET)

Exclusion Criteria:

* Atypical or psychotic subtypes of major depressive disorder.
* Alcohol or substance dependence within 12 months; abuse within 6 months, excluding nicotine Current suicidal ideations, plan or intent for self-harm; in past 3 years, repeated suicide attempts, resulting in emergency room or inpatient care.
* Major medical illness, cardiac pacemaker/defibrillator, and other implanted stimulator.
* Likely to relocate or move to a location distant from the study site within one year of enrollment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2002-06; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression, 24-item version (HRSD-24)
Clinical Global Impression (CGI) of Severity/Improvement
Psychiatric assessments will be performed every two weeks in the clinic. Once final stimulation parameters are established, psychiatric symptoms will be monitored monthly.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, MD, Principal Investigator — University Health Network, Toronto; Sidney H Kennedy, MD, FRCPC, Principal Investigator — Univesity Health Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Result] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841